CLINICAL TRIAL: NCT03287934
Title: Accuracy of Selective Laser Sintered Computer Guided Stents Versus Digital Light Processing Stents in Immediate Implant Placement in Esthetic Zone, a Randomized Controlled Study
Brief Title: Accuracy of Selective Laser Sinteredcomputer Guided Stents Versus Digital Light Processing Stents
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mahetab hamdi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.prosthodontic department
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Immediate Dental Implants
Keywords: selective laser sintering, digital light processing stents

STUDY DESIGN:
Who Masked: Participant
Masking Description: due to the nature of study only the participants could be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital light processing stent (Experimental): according to the allocation, the experimental group will receive a digital light processing stent for immediate implant drilling and placement after atraumatic extraction of the target tooth.
  Interventions: Device: selective laser sintered stent; Device: digital light processing(dlp)
- selective laser sintering (Active Comparator): according to the allocation, the intervention for the control group will be a selective laser sintering stent after atraumatic extraction of the target tooth for immediately implant placement. the selective laser sintering stent will be adapted and drilling will be done through the stent.
  Interventions: Device: selective laser sintered stent; Device: digital light processing(dlp)

INTERVENTIONS:
Device: selective laser sintered stent — after planning and virtual implant placement, a guide will be designed and the STL file will be send to prototyping center for printing the guide with selective laser sintering technique. during the surgical procedure , the target tooth will be atraumatic extracted, the stent is adapted in its place then implant drilling and placement will be done.
  Other Names: Mega selective laser sintering (brand name )
Device: digital light processing(dlp) — after planning and virtual implant placement, a guide will be designed and the STL file will be send to prototyping center for printing the guide with digital light processing technique. during the surgical procedure , the target tooth will be atraumatic extracted, the stent is adapted in its place then implant drilling and placement will be done.
  Other Names: mogassam (brand name)

SUMMARY:
patient with non-restorable tooth in the esthetic zone will be recruited in the study. a traumatic is done and implant will be placed using either digital light processed guides for control group or selective laser sintering group for intervention group.

DETAILED DESCRIPTION:
the principle investigator will randomize and equally distribute the Eligible patients between the selective laser sintering group (intervention group) and digital light processing group (control group).

* Diagnostic phase : for initial diagnosis, principle investigator will make primary impression , bite registration, face bow record and periapical x-ray for each eligible patients. The tooth to be extracted will be removed from the cast and replaced with an artificial tooth. For construction of radio graphic stent, a clear thermoplastic sheet will be pressed on the modified cast using a vacuum forming machine . A hole is done in the center of the artificial tooth packed with heated gutta percha (radiopaque material) for easy visualization on the cone beam during virtual implant placing. A dual scan protocol with cone beam CT will be made. The first scan is for the patient wearing the scan appliance while the second will be for the cast with the scan appliance.
* Planning phase : placing of the virtual implant and designing of the surgical stent will be done by virtual planning software .
* Construction of the surgical guide: principle investigator will send the Standard Language transformation (STL) file of the designed guide to a rapid prototyping center. Selective laser sintering and digital light procesing will be used for intervention and control group respectively. principle investigator will check for adaption of the guide on the cast and cement the metallic sleeve to prevent rotation during surgery.
* Surgical phase : principle investigator will prescribe a prophylactic antibiotic to the patient three days prior the surgery. Atraumatic extraction will be carried by periotomes and lancet. The integrity of the socket will be examined well by probe. The guide is stabilized in its place then drilling and implant placement will be done. Healing abutment is screwed in place to allow proper healing of the soft tissue. Patient will be instructed to avoid hard foods and follow restrict oral hygiene measures. Patient will be recalled after one week for postoperative inspection and assessment. A cone beam CT will be taken for deviation assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age should be more than 18 years old
2. Hopeless tooth in esthetic zone due to caries, endodontical problem or trauma with both neighboring teeth present.
3. Good oral hygiene
4. No periapical lesions (acute accesses or chronic fistula)
5. Adequate bone (5 mm) below the tooth to allow primary implant stability
6. Sufficient Medio-distal bone about 1.5 from each side
7. sufficient labial bone
8. sufficient band of keratinized mucosa

Exclusion Criteria:

1. heavy smoking
2. any systemic condition that is considered absolute contraindication for implant placement
3. pregnancy
4. in adequate inter-arch space
5. parafunctional habits as bruxism

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
evaluation of accuracy of implant placement clinical observation | 1 week
  measuring both angular and linear deviation of implants by virtual ruler in terms of mm

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Manil, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abduo, J., Lyons, K. & Bennamoun, M., 2014. Trends in Computer-Aided Manufacturing in Prosthodontics: A Review of the Available Streams. International Journal of Dentistry, 2014, pp.1-15. Available at: http://www.hindawi.com/journals/ijd/2014/783948/. Alzoubi, Fawaz, Nima Massoomi, and A.N., 2016. Accuracy Assessment of Immediate and Delayed Implant Placements Using CAD/CAM Surgical Guides. Journal of Oral Implantology ., 42(5), pp.391-398. Arısan, V. et al., 2013. Implant Positioning Errors in Freehand and Computer-Aided Placement Methods: A Single-Blind Clinical Comparative Study. The International Journal of Oral & Maxillofacial Implants, 28(1), pp.190-204. Available at: http://www.quintpub.com/journals/find_article.php?doi=10.11607/jomi.2691.